CLINICAL TRIAL: NCT06376877
Title: A Novel TMS Target for Anxiety: a Confirmatory Randomized Clinical Trial
Brief Title: Connectomic Targeted TMS Target for Refractory Anxiety
Acronym: ConTRA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shan Siddiqi, MD, Assistant Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P000900
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Anxiety Disorders; Mental Disorder; Psychiatric Disorder
Keywords: Transcranial Magnetic Stimulation; accelerated intermittent theta burst stimulation; theta burst stimulation; brain stimulation; neuromodulation; anxiety; transcranial; TMS; neuronavigation; neuroimaging
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Nonresponders may have the option for open label active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real aiTBS (Active Comparator): Participants in this group will receive aiTBS with neuronavigation to the anxiosomatic treatment target.
  Interventions: Procedure: Transcranial magnetic stimulation
- Sham aiTBS (Sham Comparator): Participants in this group will receive sham aiTBS with neuronavigation to the anxiosomatic treatment target.
  Interventions: Procedure: Sham transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a focal, non-invasive form of brain stimulation that has FDA clearance for depression. In this study, a form of TMS called accelerated intermittent theta burst stimulation will be administered under the supervision of a physician with TMS expertise.
  Arms: Real aiTBS
Procedure: Sham transcranial magnetic stimulation — The sham TMS coil mimics the scalp sensation of real TMS by delivering a small amount of electrical current with a pair of surface electrodes.
  Arms: Sham aiTBS

SUMMARY:
We will perform a randomized sham-controlled trial of aiTBS to an anxiosomatic circuit in patients with anxiety-related disorders (i.e., panic disorder, generalized anxiety disorder, social anxiety disorder, obsessive-compulsive disorder, and post-traumatic stress disorder). 80 participants with an anxiety-related disorder (defined below) will receive 50 active or sham TMS treatments over 5 days (following the SAINT protocol, which is FDA-cleared for MDD. The primary outcome will be the BAI, with a modified recall window to reflect the short treatment interval. Participants randomized to sham will be offered an open-label crossover extension.

DETAILED DESCRIPTION:
We recently derived a novel TMS target for anxiety via lesion and brain stimulation mapping methods. We prospectively tested this target in a sample of participants with major depressive disorder (MDD) with comorbid anxiety symptoms and found that it was more effective for anxiety (median change 60.0% vs 39.8%, p=0.01) than the conventional TMS target for MDD with comorbid anxiety. While these results are promising, it remains unclear how our target works for anxiety-related disorders as opposed to MDD comorbid anxiety symptoms. Furthermore, we used conventional 10 Hz TMS, but accelerated intermittent theta burst stimulation (aiTBS) has now been shown to improve outcomes and is now an FDA approved treatment protocol. Finally, we tested the translational hypothesis that stimulating different circuits can modify different behaviors; clinical efficacy was a secondary outcome.

This double-blinded, randomized, sham-controlled aiTBS trial will test the efficacy of our novel anxiety target. 80 participants with anxiety-related disorders (i.e., panic disorder, generalized anxiety disorder, social anxiety disorder, obsessive-compulsive disorder, and post-traumatic stress disorder) will receive 50 active or sham TMS treatments over 5 days. Changes in anxiety symptoms/processes will be assessed via validated measures (primary outcome measure: Beck Anxiety Inventory) during treatment and follow-up visits up to one-year post-treatment. Participants randomized to sham who do not respond will be offered an open-label crossover extension.

ELIGIBILITY:
Inclusion Criteria:

* English proficiency sufficient for informed consent, questionnaires/tasks, and treatment
* Diagnosis of one of the following anxiety-related disorders per Quick-SCID:

  * Generalized Anxiety Disorder
  * Social Anxiety Disorder
  * Panic Disorder
  * Posttraumatic Stress Disorder
  * Obsessive Compulsive Disorder
* Moderate level of anxiety (BAI >16)
* One failed psychological or pharmacological treatment
* Stable psychiatric medication regimen for 4 weeks prior to treatment and throughout treatment
* Primary clinician (e.g. psychiatrist, psychologist, therapist, APRN, PA, etc.) responsible for psychiatric care before, during, and after the trial
* Agreement to abstaining from becoming pregnant from screening to two weeks after treatment (the MRI visit)

Exclusion Criteria:

* • Active pregnancy as determined by a urine pregnancy test

  * Recent (within 4 weeks) or concurrent use of rapid acting antidepressant agent (ketamine/esketamine/ECT)
  * History of:

    * Exposure to TMS within the last 3 months
    * Neurosurgical intervention for psychiatric disorders
    * Autism spectrum disorder, intellectual disability, or cognitive impairment that impairs capacity to consent
    * Significant neurological illness deemed to increase risk from treatment
    * Moderate to severe neurodegenerative disease
    * Untreated or insufficiently treated endocrine disorder
    * Treatment with investigational drug or intervention during the study period
    * Bipolar I disorder or schizophrenia
  * Anyone presenting with:

    * Mania or hypomania
    * Psychosis
    * Active suicidal ideation with intent and a plan (defined by Columbia Suicide Severity Rating Scale)
    * Contraindications to either TMS or MRI (e.g., metallic implants, severe insomnia > 4 hours per night with hypnotic, etc.).
    * Current moderate or severe substance use disorder (excluding cannabis or nicotine) or demonstrating signs of acute substance withdrawal
  * Positive urine drug screen for illicit substances for cocaine, amphetamines, phencyclidine, and opioids, except for prescribed medications or known medications with history of resulting in a false positive
  * Existing tinnitus (ringing in the ears)
  * Any other condition deemed by the PI to interfere with the study or increase risk to the participant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | One week and one month after treatment
  21 item self-report scale that assesses anxiety symptoms, with a particular emphasis on physiological anxiety symptoms

SECONDARY OUTCOMES:
Inventory of Depression and Anxiety Symptoms-II | One week and one month after treatment
  99 item self-report scale of mood (e.g. dysphoria, suicidality, mania) and anxiety (e.g. social anxiety, panic, checking/ordering, traumatic avoidance/intrusion)
Hierarchical Taxonomy of Psychopathology (HiTOP)-Self Report, Distress, Fear, and Mania subfactors | One week and one month after treatment
  HiTOP is a psychiatric nosology that organizes dimensional constructs across multiple levels of abstraction (from broad spectra to specific symptoms). The HiTOP-self report Distress, Fear, and Mania subfactors contain 117 items that capture a broad range of specific mood and anxiety-relevant symptoms
State-Trait Anxiety Inventory | One week and one month after treatment
  40 item self-report scale of present anxiety (i.e., state anxiety) and the general tendency toward anxiety
Penn State Worry Questionnaire (PSWQ) | One week and one month after treatment
  16 item self-report scale of trait worry and anxious apprehension, a transdiagnostic construct characterized by a persistent pattern of negative future thinking
Mood/Anxiety Symptoms Questionnaire: Anxious Arousal (MASQ:AA) | One week and one month after treatment
  90 item self-report with a 17 item scale that measures anxious arousal, a transdiagnostic construct characterized by a persistent pattern of hyperarousal/hypervigilance
Anxiety Sensitivity Index (ASI) | One week and one month after treatment
  16 item self-report scale of concern about anxious cognitions/physiological sensations
Intolerance of Uncertainty Scale (IUS) | One week and one month after treatment
  27 item self-report scale that measures cognitive, emotional, and behavioral reactions to the potential occurrence and unpredictability of negative future events
Beck Depression Inventory (BDI) | One week and one month after treatment
  21 item self-report scale that assesses depression symptoms
TCI-R140 (Temperament and character inventory, revised 140-question format) | One week and one month after treatment
  Psychobiologically-based personality inventory which measures seven personality dimensions (harm avoidance, novelty seeking, reward dependence, persistence, self-directedness, cooperativeness, and persistence). For each dimension, this yields a scaled T-score (mean score of 50 with standard deviation of 10). This is an overall estimate of personality traits, and there are no "better" or "worse" traits.
Emotional Conflict Resolution Task | One week after treatment
  Computer task measuring accuracy and reaction time
Laboratory Fear Extinction Paradigm | One week after treatment
  We will use a validated fear extinction task (24) to assess the effects of anxiosomatic circuit TMS on fear discrimination and fear extinction. This task will consist of two learning phases: fear conditioning and fear extinction. We will measure fear via the skin conductance response.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Siddiqi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Emma Jones, Boston, Massachusetts, United States